CLINICAL TRIAL: NCT05699161
Title: Treatment of Parkinson Disease With Transplantation of SVF Cells of Adipose Origin: Safety and Exploratory Efficacy Study
Brief Title: Adipose-derived Stromal Vascular Fraction Cells to Treat Parkinson
Acronym: SVFP1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samuel Vilchez, PhD (Other)
Collaborators: Wake Forest University (Other); Ministerio de Salud, Nicaragua (Unknown); GID BIO, Inc. (Industry); National Autonomous University of Nicaragua (Other)
Responsible Party: Sponsor-Investigator, Samuel Vilchez, PhD, Professor, National Autonomous University of Nicaragua
Organization: National Autonomous University of Nicaragua (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nica-Parkinson-2021
Record Dates: First submitted 2022-12-07; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Idiopathic Parkinson Disease; Parkinson's Disease and Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group assignment. (Experimental): Bilateral treatment.
  Subdermal plane injection of SVF cells into the submuscular aponeurotic fascia of the face.
  Interventions: Genetic: Adipose-derived stromal vascular fraction cells

INTERVENTIONS:
Genetic: Adipose-derived stromal vascular fraction cells — Published minimal clinically important differences (MCID) for PDQ-39; MDS-UPDRS; and levo-dopa equivalent dose and changes in the levels of blood proteins (L-1beta, IL-2, IL-6, IL-10, and TNF-alpha) in 10 patients after 12 months of treatment with SVF cells.

SUMMARY:
This is an interventional study to treat 10 patients with a diagnosis of Parkinson's disease with neurological assessment from the Oxford Parkinson's Disease Quotient-39 (PDQ-39) and Movement Disorders Society Universal Parkinson's Disease Rating Scale (MDS-UPDRS), with autologous adipose tissue-derived stromal vascular fraction (SVF) cells by subdermal plane injection into the submuscular aponeurotic fascia of the face.

This study assesses: 1) safety and 2) feasibility and 3) exploratory evidence of efficacy.

DETAILED DESCRIPTION:
Pre-procedure/intervention evaluation

Patients had a medical history, physical exam, and medication review. Neurological examination used two instruments: PDQ-39 and the MDS-UPDRS, the latter including videorecording of a standardized motor examination. Subjects also completed the general health questionnaire SF-36 and have blood drawn for subsequent biomarker analysis (immune markers L-1beta, IL-2, IL-6, IL-10, and TNF-alpha). Patients had pre-operative laboratory studies (hemogram, coagulation profile, electrolytes, BUN, creatinine, and urinalysis) and anesthesia evaluation carried out 48 hours prior to procedures.

Surgical and biochemical technique

The autologous fat tissue was harvested via liposuction by a plastic surgeon. The fat was washed and processed with collagenase for 60 minutes at a temperature of 39-41ºC, in an incubator and by constant shaking with a rotary shaker. The digested adipose tissue was then centrifuged for 14 minutes in 3 steps and the cell fraction (SVF) contained in the fat was removed with a syringe. The cell count was performed using a Luna Stem cell counter (Logos Bio). SVF was injected the same day as the liposuction and adipose processing.

A standardized total dose of 30x10e6 SVF cells was administered [Carstens 2017]. Injections of SVF cells bilateral (into the subdermal plane along the submuscular aponeurotic fascia) 1 cc per site for a final dose of 0.3 million cells per site

Post-surgical and management of complications

Patients were observed for potentially adverse effects for 24 hours after the procedure. There were follow-up visits at seven days, 1-, 3-, 6- and 12 months postoperative and treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with UK brain bank criteria for idiopathic Parkinson's disease for a period of not less than one year
* Age 18 - 80; male or female
* Stable PD medication for at least 30 days prior to study enrollment
* A MDS-UPDRS total score > 20 and < 50
* Ability to understand the study and sign consent forms
* Intent to comply with all postoperative appointments
* Social support to be able to comply with all follow-up visits

Exclusion Criteria:

* Previous neurological disease or previous brain trauma as a confounding factor
* Cardiovascular disease or any condition that prohibits general anesthesia
* Inability to understand and / or cooperate with investigators
* Subjects that have a history of injury, infection, or deformity of at or near the anatomical site for planned product injection which may increase their risk for infection, injury, or complication related to the product (e.g., prior injury to blood vessels, lymphatics, history of orbital injury/fracture).
* Rash or possible skin infection over surgical sites or face.
* Subjects that use any form of tobacco, including e-cigarettes, more than once a week over the past year.
* Current substance abuse (drugs or alcohol) within the 6 months prior to study enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events | 12-months follow-up post intervention.
  Documentation of adverse events
L-dopa medication | Up to month 12 post intervention.
  Changes in L-dopa medication measured as levodopa-equivalent dose.
Minimal clinically important differences (MCIDs)-1 | Up to 12-months post SVF treatment
  Estimation of MCIDs scores (0-199) based on the UPDRS scale: : MCID 4.3 points low, MCID 8.1 points medium, and MCID 17.1 points high.
Minimal clinically important differences (MCIDs)-2 | Up to 12-months post SVF treatment
  Estimation of MCIDs scores (0-100) based on the PDQ-39 scale: : MCID 4.7 minimal, MCID 7.7 moderate, and MCID 10.1 significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Escuela Oscar Danilo Rosales Arguello, León, León Department, Nicaragua

REFERENCES:
- [Background] Carstens M, Haq I, Martinez-Cerrato J, Dos-Anjos S, Bertram K, Correa D. Sustained clinical improvement of Parkinson's disease in two patients with facially-transplanted adipose-derived stromal vascular fraction cells. J Clin Neurosci. 2020 Nov;81:47-51. doi: 10.1016/j.jocn.2020.09.001. Epub 2020 Sep 25. PMID 33222965
- [Background] Brown JC, Shang H, Li Y, Yang N, Patel N, Katz AJ. Isolation of Adipose-Derived Stromal Vascular Fraction Cells Using a Novel Point-of-Care Device: Cell Characterization and Review of the Literature. Tissue Eng Part C Methods. 2017 Mar;23(3):125-135. doi: 10.1089/ten.TEC.2016.0377. PMID 28177263
- [Background] Nguyen A, Guo J, Banyard DA, Fadavi D, Toranto JD, Wirth GA, Paydar KZ, Evans GR, Widgerow AD. Stromal vascular fraction: A regenerative reality? Part 1: Current concepts and review of the literature. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):170-9. doi: 10.1016/j.bjps.2015.10.015. Epub 2015 Oct 31. PMID 26565755
- [Background] Guo J, Nguyen A, Banyard DA, Fadavi D, Toranto JD, Wirth GA, Paydar KZ, Evans GR, Widgerow AD. Stromal vascular fraction: A regenerative reality? Part 2: Mechanisms of regenerative action. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):180-8. doi: 10.1016/j.bjps.2015.10.014. Epub 2015 Oct 24. PMID 26546112
- [Background] Lindvall O. Treatment of Parkinson's disease using cell transplantation. Philos Trans R Soc Lond B Biol Sci. 2015 Oct 19;370(1680):20140370. doi: 10.1098/rstb.2014.0370. PMID 26416681
- [Background] Shulman LM, Gruber-Baldini AL, Anderson KE, Fishman PS, Reich SG, Weiner WJ. The clinically important difference on the unified Parkinson's disease rating scale. Arch Neurol. 2010 Jan;67(1):64-70. doi: 10.1001/archneurol.2009.295. PMID 20065131
- [Background] Horvath K, Aschermann Z, Kovacs M, Makkos A, Harmat M, Janszky J, Komoly S, Karadi K, Kovacs N. Changes in Quality of Life in Parkinson's Disease: How Large Must They Be to Be Relevant? Neuroepidemiology. 2017;48(1-2):1-8. doi: 10.1159/000455863. Epub 2017 Feb 4. PMID 28161701